CLINICAL TRIAL: NCT05931497
Title: A Pilot Study of Whole Body Hyperthermia for Long Covid or Post-Acute Sequelae of COVID-19 (PASC)
Brief Title: Sauna for Long Covid
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Principal Investigator, Maren Nyer, Clinical Psychologist, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2023p000852
Record Dates: First submitted 2023-06-30; First posted 2023-07-05 (Actual); Last update posted 2025-11-13 (Actual); Status verified 2025-11

CONDITIONS: Long COVID
MeSH Terms: conditions — Post-Acute COVID-19 Syndrome

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized to one of two WBH groups.
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- verum whole body hyperthermia (Experimental): WBH will be completed with a Clearlight Sauna Dome and ancillary equipment to monitor core body temperature. For the verum WBH, participants will be brought to a core body temperature of 101.3°F.
  Interventions: Device: whole body hyperthermia
- sham whole body hyperthermia (Sham Comparator): The sham condition will be identical to the active WBH condition. Time and other procedures will be consistent. Mild heat will be used to mimic an active WBH session.
  Interventions: Device: whole body hyperthermia

INTERVENTIONS:
Device: whole body hyperthermia — heat will be applied to the participant through a sauna to increase core body temperature

SUMMARY:
Research suggests that Whole Body Hyperthermia in a sauna-like environment can reduce symptoms related to post-acute sequelae of SARS-CoV-2 (PASC), or Long Covid. The investigators aim to study the feasibility and treatment effect of this procedure for patients experiencing Long Covid symptoms.

DETAILED DESCRIPTION:
This proposed trial will examine, for the first-time, study whole-body hyperthermia (WBH) as a treatment for PASC. The investigators will enroll 21 people with PASC who will be randomized into two conditions with different temperature WBH. The primary aims will explore acceptability and feasibility, reduction of fatigue (primary symptom), and potential mechanisms (inflammation and sleep). Inflammation and sleep have both been shown to be dysregulated in PASC and addressed by WBH in other populations. The investigators will use week 2 as the primary endpoint. However, patients will be followed for 4 and 6 weeks to monitor the duration of effect.

ELIGIBILITY:
Inclusion Criteria:

1. 18-65 years of age
2. English language proficiency
3. Ability to provide informed consent
4. Ability to lie supine (on back) for 2 hours (required for sauna sessions)
5. Must have had clinically suspected COVID-19 and a positive antibody test or a documented SARS-CoV-2 infection (a positive reverse transcription polymerase chain reaction test) at least 12 weeks prior to Screening (Note: clinician judgment can override lack of positive COVID test with clear Long Covid onset and presentation)
6. The Patient Reported Outcome Measurement Information System Fatigue-Short Form v1.0 -Fatigue 7a (PROMIS F-SF43) raw score of 21 or greater at Screening (onset of fatigue confirmed post-infection as in other studies of PASC)
7. Individuals of childbearing potential must use an acceptable form of birth control.

Exclusion Criteria:

1. Fatigue for known reasons other than PASC (e.g. longstanding diagnosis of Chronic Fatigue Syndrome pre-dating Long Covid, low thyroid, multiple sclerosis, AIDS related fatigue, mononucleosis), as determined by clinical discretion of study investigators
2. Known hypersensitivity to infrared heat exposure, significant history of heat stroke
3. Breastfeeding, pregnancy or planned pregnancy during study
4. Active suicidal intent
5. History of bipolar disorder, psychotic disorders, eating disorders, obsessive compulsive disorder, and/or substance use or dependence (within the last year), as per the Mini-International Neuropsychiatric Interview (MINI)44
6. Positive urine toxicology screen for illicit drug use
7. Any serious unstable medical condition
8. Inability to fit into the sauna device. Morbid obesity (BMI > 40) and/or body shape that might increase the risk of cutaneous burning from the device (because of skin being too close to the heat).
9. Back pain that would interfere with ability to lay on hard surface
10. Using medication that might impact thermoregulatory capacity and cannot be held for an appropriate length (at least one half-life) as determined by clinician judgment prior to receiving WBH treatment
11. Breast Implants
12. Claustrophobia that would interfere with ability to remain in sauna
13. Unsafe cardiac status as defined by abnormal ECG reading at screening visit or as determined by study doctor or subject's physician
14. History of or current diagnosis of thrombosis or thrombophilia
15. History of hemophilia
16. History of febrile seizures or seizure disorders
17. Any new treatments/medications for long-COVID that have started in the past 3 months
18. A subject who in the opinion of the Principal Investigator would not be able to safely complete the study or would jeopardize study integrity.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2026-08-01 (Estimated); Primary Completion 2026-09-30 (Estimated); Study Completion 2026-12-01 (Estimated)

PRIMARY OUTCOMES:
The Patient Reported Outcome Measurement Information System Fatigue-Short Form v1.0 -Fatigue 7a (PROMIS F-SF) | 2-weeks (primary endpoint) follow up at 6 weeks
  provides a more in depth assessment of fatigue as compared to the PROMIS 29 and consists of 7 items that measure both the experience of fatigue and the interference of fatigue on daily activities over the past week. Uses a range of 7-35, higher scores indicate higher fatigue.

SECONDARY OUTCOMES:
Patient-Reported Outcomes Measurement Information System (PROMIS-29) | 2-weeks (primary endpoint) follow up at 6 weeks
  assesses seven health domains (i.e., physical function, fatigue, pain interference, depressive symptoms, anxiety, ability to participate in social roles and activities, and sleep disturbance) using four items per domain. There is no total score, and scores range from 4-10 for each health domain (with 4 items for each of the 7 health domains). Scores are transformed into t scores with higher scores indicating better health.
Patient Health Questionnaire-9 (PHQ) | 2-weeks (primary endpoint) follow up at 6 weeks
  a well-established, brief self-administered 9-item depression screening and monitoring tool. Uses a range of 0-27 with higher scores indicating greater depressive symptoms.
The Perceived Stress Scale (PSS) | 2-weeks (primary endpoint) follow up at 6 weeks
  consists of 10 items and measures the frequency with which perceived stressful life situations are experienced. Scores can range from 0 to 40 with higher scores indicating higher perceived stress.
Patient-Reported Outcomes Measurement Information System Cognitive Abilities | 2-weeks (primary endpoint) follow up at 6 weeks
  items target positive self-assessments of cognitive functioning with a total of 8 items. Raw scores can range from 8 to 40. The raw score is then converted to a t-score and higher scores indicate better perceived cognitive functioning.
Patient-Reported Outcomes Measurement Information System Cognitive Concerns | 2-weeks (primary endpoint) follow up at 6 weeks
  items are worded negatively and express concerns in the same areas as in the Patient-Reported Outcomes Measurement Information System Cognitive Abilities with a total of 8 items. Raw scores can range from 8 to 40. The raw score is then converted to a t-score and higher scores indicate greater cognitive concerns.
Positive and Negative Affective Schedule (PANAS) | 2-weeks (primary endpoint) follow up at 6 weeks
  consists of two 10-item mood scales to measure positive and negative affect. Raw scores range from 10 to 50. Higher scores indicate more of a positive affect.
The Composite Autonomic Symptom Score (COMPASS-31) | 2-weeks (primary endpoint) follow up at 6 weeks
  consists of 31 items and measures autonomic and neurodegenerative system symptoms. Total scores range from 0 to 100 with greater scores indicating greater autonomic dysfunction.
The Functional Assessment of Chronic Illness Therapy Fatigue Scale (FACIT-F) | 2-weeks (primary endpoint) follow up at 6 weeks
  13-item questionnaire designed to assess the severity of fatigue and its impact on daily functioning and quality of life. Respondents rate items on a 5-point scale, with higher scores indicating less fatigue. Total scores can range between 0 and 52.
Long-COVID Symptom Tool (Long-COVID ST) | 2-weeks (primary endpoint) follow up at 6 weeks
  assess the symptoms of long COVID-19 created from patients' lived experience that measures 10 different physiological domains. Scores can range from 0 to 53 with higher scores indicating greater severity of symptoms.
Long-COVID Impact Tool (Long-COVID IT) | 2-weeks (primary endpoint) follow up at 6 weeks
  assess the symptoms of long COVID-19 created from patients' lived experience that measures 10 different physiological domains. The scale also measures the impact from these symptoms. Scores can range from 0 to 60 with higher scores indicating greater life impact.

CONTACTS AND LOCATIONS:
Locations (1):
- Depression Clinical and Research Program, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No